CLINICAL TRIAL: NCT05428371
Title: A Novel, Multimodal, Machine-learning Grounded Approach to Assess the Oncological Risk of Indeterminate Thyroid Nodules
Brief Title: Assessment the Cancer Risk of Indeterminate Thyroid Nodules Through Integration of Clinical, Ultrasonographic and Multiomic Features
Acronym: THYOMICS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: Prof. Pietro Giorgio Calò (Unknown); Dott. Gian Luigi Canu (Unknown)
Responsible Party: Principal Investigator, Fabio Medas, Associate Professor, University of Cagliari
Other Study IDs: THYOMICS
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Nodule; Thyroid Cancer
Keywords: Thyroid carcinoma; Indeterminate thyroid nodule; Genomics; Proteomics; Metabolomics
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid carcinoma: Patients with indeterminate thyroid nodule and pathological diagnosis of thyroid carcinoma
  Interventions: Diagnostic Test: Multiomic analyses of blood and surgical specimens
- Follicular adenoma: Patients with indeterminate thyroid nodule and pathological diagnosis of follicular adenoma
  Interventions: Diagnostic Test: Multiomic analyses of blood and surgical specimens

INTERVENTIONS:
Diagnostic Test: Multiomic analyses of blood and surgical specimens — The following items will be evaluated:
  * cell free dna length and integrity
  * presence or absence of SNPs in cfDNA and in DNA extracted from surgical samples
  * qualitative and quantitative evaluation of serum and surgical specimens proteome (proteomics)

SUMMARY:
Indeterminate thyroid nodules have a mild risk of malignancy (15-30%). The aim of our study is to individuate new biomarkers of thyroid carcinoma through multiomic analyses of blood samples and of specimen samples of patients with indeterminate thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indeterminate thyroid nodules (Class III and Class IV according to Bethesda Classification of thyroid nodules)

Exclusion Criteria:

* Patients with concomitant thyroid nodules of Bethesda Class V or Class VI
* Patients with preoperative diagnosis of lymph node metastases of central or lateral neck compartment
* Patients with distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include in our study patients with indeterminate thyroid nodules (Class III and Class IV according to Bethesda classification) who have a mild risk of thyroid cancer (15-30%)
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers of thyroid carcinoma | 50 months
  Identification of alterations in cfDNA length and integrity, presence of SNPs in cfDNA, alterations of serum proteome predictive of thyroid carcinoma

SECONDARY OUTCOMES:
Elaboration of diagnostic algorithm | 60 months
  Elanoration of diagnostic algorithm predictive of thyroid carcinoma through integration of clinical, ultrasonographic and multiomic variables able to predict che condition of thyroid cancer in patients with indeterminate thryoid nodules

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available under reasonable request